CLINICAL TRIAL: NCT03855254
Title: Psychological Context Effects of Participant Expectation on Pain Pressure Thresholds Following Cervicothoracic HVLA Thrust Manipulation: A Double Blind, Crossover, Randomised Controlled Trial
Brief Title: Psychological Context Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Responsible Party: Principal Investigator, Darren Edwards, Principle Investigator, Swansea University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: SwanseaU1
Record Dates: First submitted 2019-02-21; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Positive Communication (Primary); Negative Communication; Control Condition
Keywords: Contextual effects

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Positive communication (Experimental)
  Interventions: Behavioral: communication type
- Control (neutral communication) (No Intervention)
- Negative communication (Experimental)
  Interventions: Behavioral: communication type

INTERVENTIONS:
Behavioral: communication type — Positive and negative communication types are the way that the practitioner communicates to the participant about the potential effectiveness of the osteopathic treatment. The control is a neutral communication condition.
  Other Names: Positive communication; Negative communication; Control
  Arms: Negative communication; Positive communication

SUMMARY:
This study explores how contextual effects in the fore of positive and negative communication can affect the effect of an osteopathic technique on pain pressure thresholds.

ELIGIBILITY:
Inclusion Criteria:

* Health volunteers with no forms of existing pain.

Exclusion Criteria:

* Participants with existing pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Pain pressure threshold | 6 months
  This is the degree to which the participant can tolerate pressure induced through an algometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Swansea University, Swansea, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Participant data may be sheared to other researcher on request.